CLINICAL TRIAL: NCT06861478
Title: In-Hospital Morbidity Associated With Proton Pump Inhibitors in Acute Variceal Bleeding and Chronic Liver Disease Treatment
Brief Title: PPIs and In-Hospital Morbidity in Acute Variceal Bleeding With Chronic Liver Disease
Acronym: Liver-IMPACT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, Luis Andrés González Torres, Resident, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GA24-00007
Record Dates: First submitted 2025-02-17; First posted 2025-03-06 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Morbidity
Keywords: Proton Bomb Inhibitors; Variceal Bleeding; Morbidity
MeSH Terms: interventions — Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Omeprazol 40 mg IV per day (Experimental): These patients are to receive omeprazole after randomization.
  Interventions: Drug: Omeprazol 40 mg IV
- No omeprazol (No Intervention): These patients are not to receive omeprazol after randomization.

INTERVENTIONS:
Drug: Omeprazol 40 mg IV — Daily until discharge
  Arms: Omeprazol 40 mg IV per day

SUMMARY:
With this study, the investigators pretend to describe intrahospital morbidity in patients living with cirrhosis (PLC) who present to the emergency department with variceal bleeding (VB).

This study is a longitudinal, prospective, experimental, analytical single-center clinical trial. The study will be performed in the Hospital Universitario "Jose E. González" de la Factultad de Medicina, Universidad Autónoma de Nuevo León, Monterrey, Nuevo León, México.

The studied population consists of adult-age patients with previous, recent, or new diagnoses of cirrhosis who present to the ED with VH without shock, infection, or acute or chronic disease with a <30% probability of death (CLIF-C <50). The exclusion criteria involve minor age, Acute Liver Failure (ALF), ICU patients, Hepatorenal Syndrome, sepsis or infection, and shock on admission except for hypovolemic and CLIF-C >50 points. Elimination criteria involve patients who want to discontinue treatment and patients with confounding endoscopic findings (Erosive esophagitis, peptic ulcers, duodenal ulcers, GAVE, and atrophic gastritis).

After the endoscopic intervention, the investigators will propose inclusion. After acceptance with Informed Consent, the investigators will randomize the patients to receive or not receive Omeprazole 40 mg IV per day until discharge. The primary outcome will represent several morbidity situations in these patients, including Hepatic Encephalopathy, intra-hospital infections, re-bleeding, shock, and acute kidney failure.

The secondary outcomes include the individual analysis of each component of our compound primary outcome, mortality by day 30, differences when grouping patients by Child-Pugh stratification, and comparing results in patients receiving omeprazole for more or less than 5 days.

DETAILED DESCRIPTION:
This is a prospective, randomized, and blinded study designed to assess the impact of proton pump inhibitor (PPI) use on in-hospital morbidity during acute variceal bleeding in patients with chronic liver disease. The clinical rationale emerges from ongoing debate regarding the safety and utility of acid suppression therapy in this population, particularly during hospitalization for portal hypertension-related bleeding.

Following initial stabilization and confirmation of upper gastrointestinal bleeding, patients undergo diagnostic endoscopy. Upon identification of varices or portal hypertensive gastropathy, eligible individuals are randomized to either continue omeprazole (40 mg daily) or discontinue PPI therapy. Randomization is conducted using computer software, and allocation concealment is maintained from the principal investigator.

Standard care protocols-including administration of vasoactive agents, prophylactic antibiotics, and endoscopic therapy-remain unaltered. The only experimental intervention involves PPI exposure during hospitalization. Clinical, biochemical, and radiological data are collected systematically throughout the hospital stay. In patients presenting with ascites, diagnostic paracentesis is performed as indicated. Events including infection, renal dysfunction, rebleeding, encephalopathy, and circulatory failure are monitored until discharge.

This study is being conducted at a tertiary university hospital with advanced endoscopy and critical care infrastructure. Institutional review board approval has been obtained. Written informed consent is obtained from each participant or their legal representative prior to enrollment.

ELIGIBILITY:
Inclusion Criteria

* Adult
* Cirrhosis
* Variceal Bleeding with only endoscopic findings consistent with portal hypertension complications
* Hypovolemic shock and Variceal bleeding

Exclusion Criteria:

* Shock of any type other than hypovolemic.
* No cirrhotic patients
* Patients that have Hepatic Encephalopathy at admission
* Hepatorenal syndrome
* Acute on chronic with CLIF-C >50 points
* Septic patients
* Spontaneous Bacterial Peritonitis

Elimination Criteria

* Voluntary removal of the study
* Patients with confounding endoscopic findings (Erosive esophagitis, peptic ulcers, duodenal ulcers, GAVE, and atrophic gastritis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2024-10-20 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
Morbidity | From the date of randomization until hospital discharge or death, assessed up to 13 weeks.
  The primary outcome is a composite dichotomous outcome represented by morbidity situations, including Hepatic Encephalopathy, intra-hospital infections, re-bleeding, shock, and acute kidney failure.

SECONDARY OUTCOMES:
Ocurrence of Hepatic Encefalopathy | From the date of randomization until hospital discharge or death, assessed up to 13 weeks.
  Binary outcome yes/ no
Ocurrence of Acute Kidney Injury | From the date of randomization until hospital discharge or death, assessed up to 13 weeks.
  Acute Kidney Failure binary yes/no
Ocurrence of Shock | From the date of randomization until hospital discharge or death, assessed up to 13 weeks.
  All types of shock except hypovolemic
Ocurrence of Re-bleeding | From the date of randomization until hospital discharge or death, assessed up to 13 weeks.
  Re-bleeding after endoscopic intervention
Ocurrence of any kind of Infection | From the date of randomization until hospital discharge or death, assessed up to 13 weeks.
  Infections after randomization
In-Hospital Mortality | From the date of randomization until hospital discharge or death, assessed up to 13 weeks.
  The investigators will assess Mortality during hospitalization
Omeprazol <or>5 days morbidity | From the date of randomization until hospital discharge or death, assessed up to 13 weeks.
  Patients who received more than or less than 5 days of omeprazole during hospitalization and morbidity
30 day Mortality | From the date of randomization until hospital discharge or death, assessed up to 13 weeks.
  The investigators will assess mortality by day 30, independently of admission status.
60 day Mortality | From the date of randomization until hospital discharge or death, assessed up to 13 weeks.
  The investigators will assess mortality by day 60, independently of admission status.
90 day Mortality | From the date of randomization until hospital discharge or death, assessed up to 13 weeks.
  The investigators will assess mortality by day 60, independently of admission status.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario "Jose E. González" de la Facultad de Medicina, Universidad Autónoma de Nuevo León, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
The investigators will decide after the finishing of this work